CLINICAL TRIAL: NCT07146802
Title: Towards a Personalized Medicine Approach to Psychological Treatment for Psychosis
Brief Title: Personalized Metacognitive Training for Psychosis: A Randomized Controlled Trial
Acronym: PERMEPSY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9603
Record Dates: First submitted 2025-08-01; First posted 2025-08-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical MCT (MCT) (Active Comparator): In this arm, participants will follow the standard Metacognitive Training (MCT) protocol. They will receive 10 one-hour sessions of classical MCT delivered in a group setting, following the current standard program. In addition to the sessions, participants will be given standardized homework tasks to reinforce the skills learned between sessions. This group serves as the active control in the study.
  Interventions: Behavioral: Metacognitive Training (MCT) for psychosis
- Personalized MCT (P-MCT) (Experimental): Participants in this arm will receive Personalized Metacognitive Training (P-MCT), an experimental intervention that uses a machine learning (ML) predictive platform to personalize the homework assignments. While the core MCT program remains unchanged, P-MCT customizes the homework based on individual patient profiles, specifically targeting areas where the patient is predicted to benefit the least. The goal is to enhance the effects of the standard MCT by providing personalized support through tailored exercises.
  Interventions: Behavioral: Metacognitive Training (MCT) for psychosis

INTERVENTIONS:
Behavioral: Metacognitive Training (MCT) for psychosis — MCT for psychosis is based on the theoretical foundations of the cognitive-behavioral model of schizophrenia, but it employs a somewhat different therapeutic approach. The program is comprised of ten modules targeting common cognitive errors, problem-solving biases as well as emotional problems in schizophrenia. These errors and biases may, on their own or in combination, culminate in the establishment of false beliefs to the point of delusions. The aim of the sessions is to raise the participants' awareness of these distortions and to prompt them to critically reflect on, expand upon, and change their current repertoire of problem solving. In addition to the sessions, the program includes homework tasks to reinforce the skills learned between sessions.

SUMMARY:
This study aims to compare the efficacy of classical Metacognitive Training (MCT) and personalized Metacognitive Training (P-MCT) for individuals with psychosis. MCT is a psychoeducational program derived from cognitive-behavioral therapy (CBT) that targets cognitive biases associated with psychotic symptoms. The goal is to assess which intervention is more effective to improve the overall functioning of individuals with psychosis. The study will use machine learning to personalize the treatment approach and evaluate its impact on clinical symptoms, cognitive functions, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 - 65 years of age.
* Patient affiliated to health insurance
* Inpatients and outpatients with DSM-5 diagnosis of schizophrenia spectrum disorder.
* Presence of positive symptoms at inclusion (PANSS delusions, suspiciousness or grandiosity ≥3).
* Stable condition with no expected changes in medication or symptoms during the last 3 months (information from clinical services, note that stable condition includes lack of suicidality).
* Patient providing informed consent.

Exclusion Criteria:

* Having received MCT in the previous year.
* Neurological disorder, or severe medical condition other than psychosis
* A score above 5 in the "Hostility" and the "Suspiciousness" items of the PANSS Positive subscale (to preserve group dynamics).
* Patient considered by his psychiatrist to be at serious risk of harm to self or others (e.g. previous aggressive or suicidal behaviors)
* Patient in an exclusion period defined by another research protocol
* Patient involved in another Investigational Medicinal Product trial
* Patient under guardianship (i.e. French "tutelle")
* Patients deprived of freedom because of a judicial measure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
P-MCT benefits on total psychotic symptoms | Day 0
  To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -). The subscale includes 7 items, each rated from 1 to 7, for a total score ranging from 7 to 49.
  Higher scores indicate more severe positive symptoms.
P-MCT benefits on total psychotic symptoms | Day 7
  To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -). The subscale includes 7 items, each rated from 1 to 7, for a total score ranging from 7 to 49.
  Higher scores indicate more severe positive symptoms.
P-MCT benefits on total psychotic symptoms | Day 14
  To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -). The subscale includes 7 items, each rated from 1 to 7, for a total score ranging from 7 to 49.
  Higher scores indicate more severe positive symptoms.
P-MCT benefits on total psychotic symptoms | Day 21
  To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -). The subscale includes 7 items, each rated from 1 to 7, for a total score ranging from 7 to 49.
  Higher scores indicate more severe positive symptoms.
P-MCT benefits on total psychotic symptoms | Day 28
  To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -). The subscale includes 7 items, each rated from 1 to 7, for a total score ranging from 7 to 49.
  Higher scores indicate more severe positive symptoms. symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -
P-MCT benefits on total psychotic symptoms | Day 35
  To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -). The subscale includes 7 items, each rated from 1 to 7, for a total score ranging from 7 to 49.
  Higher scores indicate more severe positive symptoms.
P-MCT benefits on total psychotic symptoms | Day 42
  To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -). The subscale includes 7 items, each rated from 1 to 7, for a total score ranging from 7 to 49.
  Higher scores indicate more severe positive symptoms.
P-MCT benefits on total psychotic symptoms | Day 49
  To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -). The subscale includes 7 items, each rated from 1 to 7, for a total score ranging from 7 to 49.
  Higher scores indicate more severe positive symptoms.
P-MCT benefits on total psychotic symptoms | Day 56
  To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -). The subscale includes 7 items, each rated from 1 to 7, for a total score ranging from 7 to 49.
  Higher scores indicate more severe positive symptoms.
P-MCT benefits on total psychotic symptoms | Day 63
  To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -). The subscale includes 7 items, each rated from 1 to 7, for a total score ranging from 7 to 49.
  Higher scores indicate more severe positive symptoms.
P-MCT benefits on total psychotic symptoms | Day 70
  To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -). The subscale includes 7 items, each rated from 1 to 7, for a total score ranging from 7 to 49.
  Higher scores indicate more severe positive symptoms.
P-MCT benefits on total psychotic symptoms | Months 6
  To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -To compare the benefits of P-MCT with classical MCT, we will compare total positive symptoms subscale score of the Positive and Negative Syndromes Scale (PANSS; Kay et al., 1987) -). The subscale includes 7 items, each rated from 1 to 7, for a total score ranging from 7 to 49.
  Higher scores indicate more severe positive symptoms.

IPD SHARING:
Plan to Share IPD: No